CLINICAL TRIAL: NCT07125664
Title: A Two-center, Randomized, Double-blind, Placebo-controlled Study of Intravenous Plasma-purified Alpha-1 Antitrypsin for Hospitalized Patients With COPD Exacerbations (AECOPD Study)
Brief Title: Intravenous Alpha-1 Antitrypsin for Hospitalized Patients With COPD Exacerbations (AECOPD Study)
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Fondazione IRCCS Policlinico San Matteo di Pavia (Other)
Responsible Party: Principal Investigator, Angelo Guido Corsico, MD, Fondazione IRCCS Policlinico San Matteo di Pavia
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: AECOPD study
Record Dates: First submitted 2025-08-08; First posted 2025-08-15 (Actual); Last update posted 2025-08-24 (Actual); Status verified 2025-08

CONDITIONS: Acute Exacerbation Chronic Obstructive Pulmonary Disease
Keywords: COPD exacerbations; Intravenous alpha-1 antitrypsin; IL-6; anti-inflammatory
MeSH Terms: interventions — alpha 1-Antitrypsin; Powders; Solvents; Solutions

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Prolastin (Experimental): Alpha1-proteinase inhibitor (human), commercially available as Prolastin
  Interventions: Biological: alpha1-proteinase inhibitor, produced from the plasma of human donors (Prolastin 1000 mg, powder and solvent for solution for infusion)
- Placebo (Placebo Comparator): 0.9% sodium chloride solution for infusion ("normal saline")
  Interventions: Drug: Placebo

INTERVENTIONS:
Biological: alpha1-proteinase inhibitor, produced from the plasma of human donors (Prolastin 1000 mg, powder and solvent for solution for infusion) — IV Prolastin administered once at 120 mg per kilogram of body weight
  Arms: Prolastin
Drug: Placebo — + IV administration of 0.9% sodium chloride
  Arms: Placebo

SUMMARY:
Intravenous augmentation therapy with purified preparations of AAT (Alpha1-antitrypsin) derived from human plasma is a well consolidated specific therapeutic option to treat the severe deficient state of AAT. Prolastin is used to restore the balance between AAT and elastases in the lung and consequently to prevent a further deterioration in the pulmonary emphysema. Recently, in patients with COVID-19, without genetically lowered AAT levels with moderate to severe ARDS, treatment with AAT was demonstrated to be safe, feasible, and biochemically efficacious as an anti-inflammatory therapeutic therapy.

The aim of the study, based on biological plausibility, is to evaluate the safety and efficacy (from a biological perspective) of the administration of intravenous plasma-purified AAT as an anti-inflammatory treatment for patients admitted to hospital because of a COPD exacerbation leading to an acute or an acute on chronic respiratory failure.

Thirty-six adult patients hospitalized because of a COPD exacerbation leading to an acute or an acute on chronic respiratory failure will be enrolled by the two sites involved in the study, the Pneumology Unit of Fondazione IRCCS Policlinico San Matteo (Pavia, Italy) and the Pneumology Unit of IRCCS Istituto Clinico Humanitas, Rozzano (Milano, Italy).

Participants will be randomized 2:1 in the active treatment group (standard treatment + IV administration of Prolastin) or in the placebo group (standard treatment+ IV administration of 0.9% sodium chloride).

To address the clinical question from a biological perspective, we will investigate the decrease in inflammatory markers in the active treated group in comparison with the placebo group.

The primary objective is to demonstrate a significant reduction in systemic inflammation by IV Prolastin administered once at 120 mg per kilogram of body weight in patients with moderate to severe AECOPD, as assessed by the change in plasma concentration of IL6 at 7 days after randomization, in the active treatment group with respect to placebo group.

Secondary outcomes are:

1. Difference in change in plasma concentration of IL-1b, IL-5, IL-8, IL-10, and soluble TNF receptor 1 (sTNFR1), CRP at 7 days after randomization.
2. Differences in AAT antielastase activity, the amount of active elastase, the AAT levels in serum at baseline and at 7 days after randomization.
3. Difference in treatment failure rate. Treatment failure is a composite endpoint of need for either NIV or CPAP or need of ETI or need of transfer to ICU or in-hospital death after randomization
4. Impact of AECOPD on overall health, daily life, and perceived well-being in patients with obstructive airways disease by the change of St. George's Respiratory Questionnaire (SGRQ) score from Day 7 to follow-up (30 days after hospital discharge).
5. Differences in type and number of AEs and SAEs in the two groups

The expected duration of subject participation is from randomization to 30 days after hospital discharge, with a follow up phone contact.

DETAILED DESCRIPTION:
COPD is the third leading cause of death in the world and it is characterized by airflow limitation, breathlessness, and exacerbations. Exacerbations are important events with a significant influence on prognosis and survival. Neutrophils, eosinophils, other inflammatory cells in the lung, as well as systemic inflammation and inflammatory biomarkers increase during exacerbations. Alpha1-antitrypsin (AAT) is an acute phase protein with antineutrophil elastase properties and several studies have demonstrated an elevation of acute phase proteins during COPD exacerbations. Intravenous augmentation therapy with purified preparations of AAT, derived from human plasma, is a well consolidated specific therapeutic option to treat the severe deficient state of AAT. In turn, the abrupt cessation of AAT augmentation therapy for patients with a hereditary deficiency of the protein results in increased systemic inflammation and subsequent progression of emphysema and COPD. Recently, in patients with COVID-19, without genetically lowered AAT levels with moderate to severe ARDS (Acute Respiratory Distress Syndrome), treatment with AAT was demonstrated to be safe, feasible, and biochemically efficacious as an anti-inflammatory therapy. This suggests a potential protective effect of AAT in treating COPD exacerbations in subjects without the genetic deficiency of AAT because of the anti-inflammatory effect of AAT.

Primary objective:

- to demonstrate a significant reduction in systemic inflammation by IV Prolastin administered once at 120 mg per kilogram of body weight in patients with moderate to severe AECOPD, as assessed by the change in plasma concentration of IL6 at 7 days after randomization, in the active treatment group with respect to placebo group.

Secondary objectives:

1. to determine the anti-inflammatory and immunomodulatory effects of IV Prolastin administered once at 120 mg per kilogram of body weight on plasma concentration of other biomarkers which have been implicated in pulmonary and systemic inflammation, and also to be suppressed by AAT in vivo
2. to identify treatment failure as assessed by:

   1. need for either NIV or CPAP
   2. need of ETI
   3. need of transfer to ICU
   4. in-hospital death after randomization
3. to evaluate the impact of AECOPD on overall health, daily life, and perceived well-being in patients with obstructive airways disease at discharge
4. to determine the safety of IV Prolastin administered once at 120 mg per kilogram of body weight, as assessed by the type and number of AEs and SAEs in the two groups.

   Primary study outcome:

   • change in level of circulating IL-6 in plasma at 7 days after IMP administration, as measured by ELISA.

   Secondary study outcomes:
   * change in plasma concentration of IL-1b, IL-5, IL-8, IL-10, and soluble TNF receptor 1(sTNFR1), CRP at 7 days after randomization
   * differences in the AAT antielastase activity, the amount of active elastase, the AAT levels in serum at baseline and at 7 days after randomization
   * treatment failure (need for either NIV or CPAP or ETI or transfer to ICU or in-hospital death after randomization)
   * differences in SGRQ score at discharge
   * differences in type and number of AEs and SAEs in the two groups.

   Recruitment will take place at the Pneumology Unit of Fondazione IRCCS Policlinico San Matteo (Pavia, Italy) and at the Pneumology Unit of IRCCS Istituto Clinico Humanitas, Rozzano (Milano, Italy), during the hospitalization because of a COPD exacerbation leading to an acute or an acute on chronic respiratory failure.

   At the Screening day, the following data will be collected: demographics (date of birth, sex, ethnicity), medical history and medications (previous and concomitant, including those administered at emergency room access), vital signs (systolic/diastolic blood pressure, heart rate, peripheral oxygen saturation, respiratory rate), electrocardiogram. The following screening assessments will be undertaken to ensure that a patient meets the criteria for enrolment:
   * chest imaging review (X-ray or CT scan performed per routine clinical practice at the hospital admission)
   * physical examination
   * confirmation of a moderate to severe ECOPD (exacerbations of COPD), according to the Rome proposal
   * sputum NEAT stik

   At the Baseline day (if different from the screening day), a physical examination will be performed and vital signs will be collected again. Before randomization, the following laboratory assessments will be carried out as per routine clinical care (blood count, basic liver/renal/bone profile biochemistry, standard markers of inflammation such as C-reactive protein, arterial blood gas analysis). A plasma sample will be obtained for cytokine measurements (IL-6, IL-1b, IL-5, IL-8, IL-10, sTNFR1), for AAT antielastase activity, active elastase ad serum AAT level before randomization. Within 24 hours by the admission to the respiratory ward, subjects who meet inclusion criteria will be randomized 2:1 to one of the two study arms (Prolastin or placebo), according to a computer-generated random blocks randomization list. Both the active drug and matching placebo will be prepared by unblinded trial personnel.

   At the Baseline day the investigational product (Prolastin or placebo) will be administered, concomitant medications will be collected and the adverse events evaluation will be performed.

   At Day 7 (seven day after IMP administration) the following assessments will be performed:
   * physical examination
   * vital signs collection (blood pressure, mean arterial pressure, heart rate, temperature, peripheral oxygen saturation, respiratory rate, where appropriate)
   * electrocardiogram
   * blood sample for CRP, ABG analysis, as per normal clinical practice
   * plasma sample collection for cytokine measurements (IL-6, IL-1b, IL-5, IL-8, IL-10, sTNFR1), for AAT antielastase activity, active elastase and serum AAT level
   * adverse events evaluation
   * concomitant medication collection
   * St. George's Respiratory Questionnaire (SGRQ) administration

   At the Hospital Discharge Day, the following data will be collected:
   * physical examination
   * vital signs (blood pressure, mean arterial pressure, heart rate, temperature, peripheral oxygen saturation, respiratory rate, where appropriate)
   * adverse events
   * concomitant medication
   * additional clinical findings occurred during the hospital stay (need for either NIV or CPAP or ETI or ICU admission and total days in ICU)

   A Phone contact, 30 days after discharge, will be done to record:
   * adverse events
   * concomitant medication
   * SGRQ responses
   * additional clinical findings after hospital discharge

ELIGIBILITY:
Inclusion Criteria:

1. Informed Consent as documented by signature
2. Male and female ≥40 years old
3. Previous COPD diagnosis with a documented post-bronchodilator FEV1 to FVC ratio (FEV1/FVC) equal to or less than 0.70 or LLN
4. Hospitalized for a moderate to severe exacerbation, according to the Rome proposal
5. Admission to the respiratory ward by ≤24 hours
6. Acute respiratory failure with SpO2 <92% at room air, or PaO2< 60 mmHg at room air, or acute on chronic respiratory failure defined as higher Increased oxygen requirements compared with the home standard oxygen prescription
7. A positive sputum NEATstik®, that corresponds to an approximate neutrophil elastase concentration of 8 μg·mL-1 (rapid point-of-care test)

Exclusion Criteria:

1. Clinically important pulmonary disease other than COPD (e.g., clinically significant bronchiectasis, pulmonary fibrosis, cystic fibrosis, hypoventilation syndrome associated with obesity, lung cancer, and primary ciliary dyskinesia)
2. Presence of pneumonia or other pleuroparenchymal abnormalities on either chest X-ray or Chest CT scan, performed per routine clinical practice at the hospital admission
3. Current diagnosis of asthma according to the GINA, prior history of asthma, or asthma-COPD overlap
4. Known AATD as homozygous or composite heterozygous mutation
5. Presence of any active malignancy (other than non-melanoma skin cancer)
6. Any unstable disorder, including, but not limited to, cardiovascular, gastrointestinal, hepatic, renal, neurological, musculoskeletal, infectious, endocrine, metabolic, haematological, psychiatric disorder, major physical and/or cognitive impairment that, in the opinion of the Investigator, could:

   1. Affect the safety of the participant throughout the study
   2. Influence the findings of the study or their interpretation
7. Known diagnosis of selective IgA deficiency defined as a serum IgA of less than 7 mg/dl (0.07 g/L)
8. Patient with the immediate need for ETI of NIV (patients already on CPAP or NIV can be included)
9. Contraindications to the class of drugs under study, e.g. known hypersensitivity or allergy to class of drugs or the investigational product
10. Women who are of childbearing potential*
11. Participants that have previously received Prolastin® 1000 mg/40 ml
12. Participation in another interventional clinical trials with investigational drugs within the 30 days preceding and during the present study. * A woman is considered of childbearing potential, i.e. fertile, following menarche and until becoming post-menopausal unless permanently sterile. Permanent sterilisation methods include hysterectomy, bilateral salpingectomy and bilateral oophorectomy. Women will be considered postmenopausal if they have been amenorrhoeic for 12 months prior to the randomisation without an alternative medical cause.

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Estimated)
Dates: Start 2025-10-01 (Estimated); Primary Completion 2027-10-07 (Estimated); Study Completion 2027-12-01 (Estimated)

PRIMARY OUTCOMES:
Change in level of circulating IL-6 in plasma | at 7 days after IMP administration
  change in level of circulating IL-6 in plasma at 7 days after IMP administration, as measured by ELISA

SECONDARY OUTCOMES:
Change in plasma concentration of IL-1b, IL-5, IL-8, IL-10, and soluble TNF receptor 1(sTNFR1), CRP | at 7 days after after randomization
  change in plasma concentration of IL-1b, IL-5, IL-8, IL-10, and soluble TNF receptor 1(sTNFR1), CRP at 7 days after randomization
Differences in the AAT antielastase activity, the amount of active elastase, the AAT levels in serum | at baseline and at 7 days after randomization
  differences in the AAT antielastase activity, the amount of active elastase, the AAT levels in serum at baseline and at 7 days after randomization
Treatment failure | from randomization to 30 days after hospital discharge
  treatment failure (need for either NIV or CPAP or ETI or transfer to ICU or in-hospital death after randomization)
Impact of AECOPD on overall health, daily life, and perceived well-being | from Day 7 to 30 days after hospital discharge
  Impact of AECOPD on overall health, daily life, and perceived well-being in patients with obstructive airways disease by the change of St. George's Respiratory Questionnaire (SGRQ) score (scores are expressed as a percentage of overall impairment where 100 represents worst possible health status and 0 indicates best possible health status) from Day 7 to follow-up (30 days after hospital discharge)
Type and number of AEs and SAEs | from randomization to 30 days after hospital discharged
  Differences in type and number of AEs and SAEs in the two groups (active and placebo)

CONTACTS AND LOCATIONS:
Locations (1):
- Fondazione IRCCS Policlinico San Matteo, Pavia, Lombardy, Italy

REFERENCES:
- [Background] Celli BR, Fabbri LM, Aaron SD, Agusti A, Brook R, Criner GJ, Franssen FME, Humbert M, Hurst JR, O'Donnell D, Pantoni L, Papi A, Rodriguez-Roisin R, Sethi S, Torres A, Vogelmeier CF, Wedzicha JA. An Updated Definition and Severity Classification of Chronic Obstructive Pulmonary Disease Exacerbations: The Rome Proposal. Am J Respir Crit Care Med. 2021 Dec 1;204(11):1251-1258. doi: 10.1164/rccm.202108-1819PP. No abstract available. PMID 34570991
- [Background] Bristow CL. Measuring the Concentration of Active Alpha-1 Antitrypsin in Serum. Methods Mol Biol. 2024;2750:71-77. doi: 10.1007/978-1-0716-3605-3_7. PMID 38108968
- [Background] Lee MC, Wu WY, Lu HY, Hsieh HN, Wu WH. Conducting the non-inferiority test for the means with unknown coefficient of variation in a three-arm trial. BMC Med Res Methodol. 2023 Aug 11;23(1):183. doi: 10.1186/s12874-023-01990-w. PMID 37568109
- [Background] Escribano Duenas AM, Martin Garcia M, Tortajada Goitia B, Arenas Villafranca JJ. Case report: Self-administration of alpha-1 antitrypsin therapy: a report of two cases. Front Pharmacol. 2023 Nov 21;14:1291677. doi: 10.3389/fphar.2023.1291677. eCollection 2023. PMID 38074132
- [Background] Blanco I, Lara B, de Serres F. Efficacy of alpha1-antitrypsin augmentation therapy in conditions other than pulmonary emphysema. Orphanet J Rare Dis. 2011 Apr 12;6:14. doi: 10.1186/1750-1172-6-14. PMID 21486454
- [Background] Wencker M, Banik N, Buhl R, Seidel R, Konietzko N. Long-term treatment of alpha1-antitrypsin deficiency-related pulmonary emphysema with human alpha1-antitrypsin. Wissenschaftliche Arbeitsgemeinschaft zur Therapie von Lungenerkrankungen (WATL)-alpha1-AT-study group. Eur Respir J. 1998 Feb;11(2):428-33. doi: 10.1183/09031936.98.11020428. PMID 9551749
- [Background] Stoller JK, Fallat R, Schluchter MD, O'Brien RG, Connor JT, Gross N, O'Neil K, Sandhaus R, Crystal RG. Augmentation therapy with alpha1-antitrypsin: patterns of use and adverse events. Chest. 2003 May;123(5):1425-34. doi: 10.1378/chest.123.5.1425. PMID 12740257
- [Background] Hubbard RC, Sellers S, Czerski D, Stephens L, Crystal RG. Biochemical efficacy and safety of monthly augmentation therapy for alpha 1-antitrypsin deficiency. JAMA. 1988 Sep 2;260(9):1259-64. PMID 3261353
- [Background] Greulich T, Chlumsky J, Wencker M, Vit O, Fries M, Chung T, Shebl A, Vogelmeier C, Chapman KR, McElvaney NG; RAPID Trial Group. Safety of biweekly alpha1-antitrypsin treatment in the RAPID programme. Eur Respir J. 2018 Nov 29;52(5):1800897. doi: 10.1183/13993003.00897-2018. Print 2018 Nov. PMID 30237305
- [Background] Murphy MP, McEnery T, McQuillan K, McElvaney OF, McElvaney OJ, Landers S, Coleman O, Bussayajirapong A, Hawkins P, Henry M, Meleady P, Reeves EP, McElvaney NG. alpha1 Antitrypsin therapy modulates the neutrophil membrane proteome and secretome. Eur Respir J. 2020 Apr 30;55(4):1901678. doi: 10.1183/13993003.01678-2019. Print 2020 Apr. PMID 32060059
- [Background] Bergin DA, Reeves EP, Meleady P, Henry M, McElvaney OJ, Carroll TP, Condron C, Chotirmall SH, Clynes M, O'Neill SJ, McElvaney NG. alpha-1 Antitrypsin regulates human neutrophil chemotaxis induced by soluble immune complexes and IL-8. J Clin Invest. 2010 Dec;120(12):4236-50. doi: 10.1172/JCI41196. Epub 2010 Nov 8. PMID 21060150
- [Background] Elliott PR, Pei XY, Dafforn TR, Lomas DA. Topography of a 2.0 A structure of alpha1-antitrypsin reveals targets for rational drug design to prevent conformational disease. Protein Sci. 2000 Jul;9(7):1274-81. doi: 10.1110/ps.9.7.1274. PMID 10933492
- [Background] Greene CM, McElvaney NG. Proteases and antiproteases in chronic neutrophilic lung disease - relevance to drug discovery. Br J Pharmacol. 2009 Oct;158(4):1048-58. doi: 10.1111/j.1476-5381.2009.00448.x. PMID 19845686
- [Background] Wewers MD, Casolaro MA, Sellers SE, Swayze SC, McPhaul KM, Wittes JT, Crystal RG. Replacement therapy for alpha 1-antitrypsin deficiency associated with emphysema. N Engl J Med. 1987 Apr 23;316(17):1055-62. doi: 10.1056/NEJM198704233161704. PMID 3494198
- [Background] McElvaney NG, Burdon J, Holmes M, Glanville A, Wark PA, Thompson PJ, Hernandez P, Chlumsky J, Teschler H, Ficker JH, Seersholm N, Altraja A, Makitaro R, Chorostowska-Wynimko J, Sanak M, Stoicescu PI, Piitulainen E, Vit O, Wencker M, Tortorici MA, Fries M, Edelman JM, Chapman KR; RAPID Extension Trial Group. Long-term efficacy and safety of alpha1 proteinase inhibitor treatment for emphysema caused by severe alpha1 antitrypsin deficiency: an open-label extension trial (RAPID-OLE). Lancet Respir Med. 2017 Jan;5(1):51-60. doi: 10.1016/S2213-2600(16)30430-1. Epub 2016 Dec 2. PMID 27916480
- [Background] Campos MA, Geraghty P, Holt G, Mendes E, Newby PR, Ma S, Luna-Diaz LV, Turino GM, Stockley RA. The Biological Effects of Double-Dose Alpha-1 Antitrypsin Augmentation Therapy. A Pilot Clinical Trial. Am J Respir Crit Care Med. 2019 Aug 1;200(3):318-326. doi: 10.1164/rccm.201901-0010OC. PMID 30965011
- [Background] McElvaney OJ, McEvoy NL, Boland F, McElvaney OF, Hogan G, Donnelly K, Friel O, Browne E, Fraughen DD, Murphy MP, Clarke J, Choileain ON, O'Connor E, McGuinness R, Boylan M, Kelly A, Hayden JC, Collins AM, Cullen A, Hyland D, Carroll TP, Geoghegan P, Laffey JG, Hennessy M, Martin-Loeches I, McElvaney NG, Curley GF. A randomized, double-blind, placebo-controlled trial of intravenous alpha-1 antitrypsin for ARDS secondary to COVID-19. Med. 2022 Apr 8;3(4):233-248.e6. doi: 10.1016/j.medj.2022.03.001. Epub 2022 Mar 11. PMID 35291694
- [Background] Chapman KR, Burdon JG, Piitulainen E, Sandhaus RA, Seersholm N, Stocks JM, Stoel BC, Huang L, Yao Z, Edelman JM, McElvaney NG; RAPID Trial Study Group. Intravenous augmentation treatment and lung density in severe alpha1 antitrypsin deficiency (RAPID): a randomised, double-blind, placebo-controlled trial. Lancet. 2015 Jul 25;386(9991):360-8. doi: 10.1016/S0140-6736(15)60860-1. Epub 2015 May 27. PMID 26026936
- [Background] Ritzmann F, Chitirala P, Kruger N, Hoffmann M, Zuo W, Lammert F, Smola S, Tov N, Alagem N, Lepper PM, Pohlmann S, Beisswenger C, Herr C, Bals R; AAT-in-COVID-19 Study Group. Therapeutic Application of Alpha-1 Antitrypsin in COVID-19. Am J Respir Crit Care Med. 2021 Jul 15;204(2):224-227. doi: 10.1164/rccm.202104-0833LE. No abstract available. PMID 33961754
- [Background] McElvaney OJ, O'Connor E, McEvoy NL, Fraughan DD, Clarke J, McElvaney OF, Gunaratnam C, O'Rourke J, Curley GF, McElvaney NG. Alpha-1 antitrypsin for cystic fibrosis complicated by severe cytokinemic COVID-19. J Cyst Fibros. 2021 Jan;20(1):31-35. doi: 10.1016/j.jcf.2020.11.012. Epub 2020 Nov 20. PMID 33288475
- [Background] Lockett AD, Kimani S, Ddungu G, Wrenger S, Tuder RM, Janciauskiene SM, Petrache I. alpha(1)-Antitrypsin modulates lung endothelial cell inflammatory responses to TNF-alpha. Am J Respir Cell Mol Biol. 2013 Jul;49(1):143-50. doi: 10.1165/rcmb.2012-0515OC. PMID 23526215
- [Background] Pott GB, Chan ED, Dinarello CA, Shapiro L. Alpha-1-antitrypsin is an endogenous inhibitor of proinflammatory cytokine production in whole blood. J Leukoc Biol. 2009 May;85(5):886-95. doi: 10.1189/jlb.0208145. Epub 2009 Feb 5. PMID 19197072
- [Background] Nita I, Hollander C, Westin U, Janciauskiene SM. Prolastin, a pharmaceutical preparation of purified human alpha1-antitrypsin, blocks endotoxin-mediated cytokine release. Respir Res. 2005 Jan 31;6(1):12. doi: 10.1186/1465-9921-6-12. PMID 15683545
- [Background] Janciauskiene S, Wrenger S, Immenschuh S, Olejnicka B, Greulich T, Welte T, Chorostowska-Wynimko J. The Multifaceted Effects of Alpha1-Antitrypsin on Neutrophil Functions. Front Pharmacol. 2018 Apr 17;9:341. doi: 10.3389/fphar.2018.00341. eCollection 2018. PMID 29719508
- [Background] Aldonyte R, Jansson L, Janciauskiene S. Concentration-dependent effects of native and polymerised alpha1-antitrypsin on primary human monocytes, in vitro. BMC Cell Biol. 2004 Mar 29;5:11. doi: 10.1186/1471-2121-5-11. PMID 15050036
- [Background] Tilg H, Vannier E, Vachino G, Dinarello CA, Mier JW. Antiinflammatory properties of hepatic acute phase proteins: preferential induction of interleukin 1 (IL-1) receptor antagonist over IL-1 beta synthesis by human peripheral blood mononuclear cells. J Exp Med. 1993 Nov 1;178(5):1629-36. doi: 10.1084/jem.178.5.1629. PMID 7693853
- [Background] Stockley RA, Bayley DL, Unsal I, Dowson LJ. The effect of augmentation therapy on bronchial inflammation in alpha1-antitrypsin deficiency. Am J Respir Crit Care Med. 2002 Jun 1;165(11):1494-8. doi: 10.1164/rccm.2109013. PMID 12045122
- [Background] Lewis EC. Expanding the clinical indications for alpha(1)-antitrypsin therapy. Mol Med. 2012 Sep 7;18(1):957-70. doi: 10.2119/molmed.2011.00196. PMID 22634722
- [Background] McCarthy C, Reeves EP, McElvaney NG. The Role of Neutrophils in Alpha-1 Antitrypsin Deficiency. Ann Am Thorac Soc. 2016 Aug;13 Suppl 4:S297-304. doi: 10.1513/AnnalsATS.201509-634KV. PMID 27564664
- [Background] Jonigk D, Al-Omari M, Maegel L, Muller M, Izykowski N, Hong J, Hong K, Kim SH, Dorsch M, Mahadeva R, Laenger F, Kreipe H, Braun A, Shahaf G, Lewis EC, Welte T, Dinarello CA, Janciauskiene S. Anti-inflammatory and immunomodulatory properties of alpha1-antitrypsin without inhibition of elastase. Proc Natl Acad Sci U S A. 2013 Sep 10;110(37):15007-12. doi: 10.1073/pnas.1309648110. Epub 2013 Aug 23. PMID 23975926
- [Background] Janciauskiene SM, Bals R, Koczulla R, Vogelmeier C, Kohnlein T, Welte T. The discovery of alpha1-antitrypsin and its role in health and disease. Respir Med. 2011 Aug;105(8):1129-39. doi: 10.1016/j.rmed.2011.02.002. Epub 2011 Mar 1. PMID 21367592
- [Background] Ingebrigtsen TS, Marott JL, Rode L, Vestbo J, Lange P, Nordestgaard BG. Fibrinogen and alpha1-antitrypsin in COPD exacerbations. Thorax. 2015 Nov;70(11):1014-21. doi: 10.1136/thoraxjnl-2015-207561. Epub 2015 Aug 24. PMID 26304913
- [Background] Dahl M, Nordestgaard BG, Lange P, Vestbo J, Tybjaerg-Hansen A. Molecular diagnosis of intermediate and severe alpha(1)-antitrypsin deficiency: MZ individuals with chronic obstructive pulmonary disease may have lower lung function than MM individuals. Clin Chem. 2001 Jan;47(1):56-62. PMID 11148177
- [Background] Turino GM, Barker AF, Brantly ML, Cohen AB, Connelly RP, Crystal RG, Eden E, Schluchter MD, Stoller JK. Clinical features of individuals with PI*SZ phenotype of alpha 1-antitrypsin deficiency. alpha 1-Antitrypsin Deficiency Registry Study Group. Am J Respir Crit Care Med. 1996 Dec;154(6 Pt 1):1718-25. doi: 10.1164/ajrccm.154.6.8970361.
- [Background] Silverman EK, Sandhaus RA. Clinical practice. Alpha1-antitrypsin deficiency. N Engl J Med. 2009 Jun 25;360(26):2749-57. doi: 10.1056/NEJMcp0900449. No abstract available. PMID 19553648
- [Background] Fregonese L, Stolk J. Hereditary alpha-1-antitrypsin deficiency and its clinical consequences. Orphanet J Rare Dis. 2008 Jun 19;3:16. doi: 10.1186/1750-1172-3-16. PMID 18565211
- [Background] Bafadhel M, McKenna S, Terry S, Mistry V, Pancholi M, Venge P, Lomas DA, Barer MR, Johnston SL, Pavord ID, Brightling CE. Blood eosinophils to direct corticosteroid treatment of exacerbations of chronic obstructive pulmonary disease: a randomized placebo-controlled trial. Am J Respir Crit Care Med. 2012 Jul 1;186(1):48-55. doi: 10.1164/rccm.201108-1553OC. Epub 2012 Mar 23. PMID 22447964
- [Background] Waljee AK, Rogers MA, Lin P, Singal AG, Stein JD, Marks RM, Ayanian JZ, Nallamothu BK. Short term use of oral corticosteroids and related harms among adults in the United States: population based cohort study. BMJ. 2017 Apr 12;357:j1415. doi: 10.1136/bmj.j1415. PMID 28404617
- [Background] Sivapalan P, Ingebrigtsen TS, Rasmussen DB, Sorensen R, Rasmussen CM, Jensen CB, Allin KH, Eklof J, Seersholm N, Vestbo J, Jensen JS. COPD exacerbations: the impact of long versus short courses of oral corticosteroids on mortality and pneumonia: nationwide data on 67 000 patients with COPD followed for 12 months. BMJ Open Respir Res. 2019 Mar 30;6(1):e000407. doi: 10.1136/bmjresp-2019-000407. eCollection 2019. PMID 31179005
- [Background] Aaron SD, Vandemheen KL, Hebert P, Dales R, Stiell IG, Ahuja J, Dickinson G, Brison R, Rowe BH, Dreyer J, Yetisir E, Cass D, Wells G. Outpatient oral prednisone after emergency treatment of chronic obstructive pulmonary disease. N Engl J Med. 2003 Jun 26;348(26):2618-25. doi: 10.1056/NEJMoa023161. PMID 12826636
- [Background] Alia I, de la Cal MA, Esteban A, Abella A, Ferrer R, Molina FJ, Torres A, Gordo F, Elizalde JJ, de Pablo R, Huete A, Anzueto A. Efficacy of corticosteroid therapy in patients with an acute exacerbation of chronic obstructive pulmonary disease receiving ventilatory support. Arch Intern Med. 2011 Nov 28;171(21):1939-46. doi: 10.1001/archinternmed.2011.530. PMID 22123804
- [Background] Thompson WH, Nielson CP, Carvalho P, Charan NB, Crowley JJ. Controlled trial of oral prednisone in outpatients with acute COPD exacerbation. Am J Respir Crit Care Med. 1996 Aug;154(2 Pt 1):407-12. doi: 10.1164/ajrccm.154.2.8756814.
- [Background] Niewoehner DE, Erbland ML. Systemic corticosteroids in COPD. An unresolved clinical dilemma. Chest. 1996 Oct;110(4):867-9. doi: 10.1378/chest.110.4.867-a. No abstract available. PMID 8874233
- [Background] Maltais F, Ostinelli J, Bourbeau J, Tonnel AB, Jacquemet N, Haddon J, Rouleau M, Boukhana M, Martinot JB, Duroux P. Comparison of nebulized budesonide and oral prednisolone with placebo in the treatment of acute exacerbations of chronic obstructive pulmonary disease: a randomized controlled trial. Am J Respir Crit Care Med. 2002 Mar 1;165(5):698-703. doi: 10.1164/ajrccm.165.5.2109093. PMID 11874817
- [Background] Davies L, Angus RM, Calverley PM. Oral corticosteroids in patients admitted to hospital with exacerbations of chronic obstructive pulmonary disease: a prospective randomised controlled trial. Lancet. 1999 Aug 7;354(9177):456-60. doi: 10.1016/s0140-6736(98)11326-0. PMID 10465169
- [Background] Groenke L, Disse B. Blood eosinophil counts as markers of response to inhaled corticosteroids in COPD? Lancet Respir Med. 2015 Aug;3(8):e26. doi: 10.1016/S2213-2600(15)00258-1. No abstract available. PMID 26282478
- [Background] Baines KJ, Pavord ID, Gibson PG. The role of biomarkers in the management of airways disease. Int J Tuberc Lung Dis. 2014 Nov;18(11):1264-8. doi: 10.5588/ijtld.14.0226. PMID 25299856
- [Background] Bafadhel M, McKenna S, Terry S, Mistry V, Reid C, Haldar P, McCormick M, Haldar K, Kebadze T, Duvoix A, Lindblad K, Patel H, Rugman P, Dodson P, Jenkins M, Saunders M, Newbold P, Green RH, Venge P, Lomas DA, Barer MR, Johnston SL, Pavord ID, Brightling CE. Acute exacerbations of chronic obstructive pulmonary disease: identification of biologic clusters and their biomarkers. Am J Respir Crit Care Med. 2011 Sep 15;184(6):662-71. doi: 10.1164/rccm.201104-0597OC. PMID 21680942
- [Background] Ingebrigtsen TS, Marott JL, Vestbo J, Hallas J, Nordestgaard BG, Dahl M, Lange P. Characteristics of undertreatment in COPD in the general population. Chest. 2013 Dec;144(6):1811-1818. doi: 10.1378/chest.13-0453. PMID 23989916
- [Background] Hurst JR, Vestbo J, Anzueto A, Locantore N, Mullerova H, Tal-Singer R, Miller B, Lomas DA, Agusti A, Macnee W, Calverley P, Rennard S, Wouters EF, Wedzicha JA; Evaluation of COPD Longitudinally to Identify Predictive Surrogate Endpoints (ECLIPSE) Investigators. Susceptibility to exacerbation in chronic obstructive pulmonary disease. N Engl J Med. 2010 Sep 16;363(12):1128-38. doi: 10.1056/NEJMoa0909883. PMID 20843247
- [Background] Venkatesan P. GOLD COPD report: 2023 update. Lancet Respir Med. 2023 Jan;11(1):18. doi: 10.1016/S2213-2600(22)00494-5. Epub 2022 Nov 30. No abstract available. PMID 36462509
- [Background] GBD 2019 Diseases and Injuries Collaborators. Global burden of 369 diseases and injuries in 204 countries and territories, 1990-2019: a systematic analysis for the Global Burden of Disease Study 2019. Lancet. 2020 Oct 17;396(10258):1204-1222. doi: 10.1016/S0140-6736(20)30925-9. PMID 33069326